CLINICAL TRIAL: NCT04023578
Title: Mobility and Perceived Functioning of Unilateral Transfemoral Amputees, Comparison of Hydraulic and Magneto-rheologic Microprocessor Controlled Knees.
Brief Title: An Investigation of Functional Improvements in the RHEO KNEE Compared to Hydraulic Microprocessor Controlled Knees (MPKs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Baker Orthotics & Prosthetics (Industry); Virginia Prosthetics & Orthotics (Industry); Methodist Rehabilitation Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-P197
Record Dates: First submitted 2019-07-16; First posted 2019-07-17 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Rheo Knee XC (Experimental): Amputee subjects currently using either magneto-rehologic or hydraulic MPKs are fitted with the Rheo Knee XC, a magneto-rheologic MPK.
  Interventions: Device: RHEO KNEE XC

INTERVENTIONS:
Device: RHEO KNEE XC — Microprocessor controlled knee using Magneto-Rheologic techonology.

SUMMARY:
The aim of this study was to evaluate the mobility, perceived safety and functioning of unilateral transfemoral (TF) amputees using the Rheo Knee XC compared to their existing prosthetic knee (RHEO KNEE II, III or Genium, X2 or X3) after 3 weeks of use.

The primary objective of the study was to determine/investigate whether unilateral (TF) amputees can apply and benefit from the stair ascent function of the Rheo Knee XC and compare the stair ascent function and automatic cycling detection of the Rheo Knee XC to hydraulic microprocessor controlled knees (MPK-HY).

The testing was conducted in a non-blinded, multicenter, prospective within subject comparison, with a subgroup analysis with Magneto-rheologic microprocessor controlled knees (MPK-MR) subgroup and MPK-HY subgroup comparing to the Rheo knee XC.

A convenience sample of 15 transfemoral amputee users was recruited at 4 study sites.

Inclusion criteria:

* Cognitive ability to understand all instructions and questionnaires in the study;
* Unilateral knee-disarticulated or transfemoral users fitted to Rheo Knee II,III or Genium
* Willing and able to participate in the study and follow the protocol
* Confident prosthetic users for more than 3 months
* Older than 18 years Exclusion Criteria
* Patients with the following characteristics are not eligible for study entry:
* 50Kg> body weight > 136Kg
* Users with cognitive impairment
* Users not understanding the function of the knee
* Users not able to charge the battery Testing was conducted between June and August 2015 in four US locations. Participants visited the study location twice, for approximately 3 hours per visit. First time for the baseline measure and initial fitting and secondly after 3 weeks of accommodation on the Rheo knee XC, performing the same measures as for the baseline. Measures included 6 minute walk test with Borg scale CR pre and post, L-test, stair assessment index, stair and bicycle evaluation and Prosthesis evaluation questionnaire mobility section (PEQ MS12/5)

For statistics repeated measures analysis of variance (ANOVA) comparing baseline to 3 week follow up were performed.

DETAILED DESCRIPTION:
Recruiting and participants:

A convenience sample of 15 transfemoral amputee users was recruited at 4 study sites. Potential subjects were identified from the customer base of study sites, local investigators evaluated , based on previous experience of interaction with and servicing of patients, if a potential participant is cognitively capable. If a potential participant fitted the inclusion and exclusion criteria the local investigator (CPO-Certified prosthetist/orthotist) contacted them via telephone. During the telephone call the investigator verified if they were interested in participating in the study. If interest was expressed and eligibility criteria was met an appointment was made for enrollment in the study. Informed consent was obtained from all participants at the beginning of the first visit, prior to clinical testing and prosthetic fitting.

Setting:

Testing was conducted in four US locations with daily mean temperature during the testing period between 79.3 to 85.3 degrees Fahrenheit, Fort Worth (Baker orthotics & prosthetics), Jackson (Methodist Rehabilitation Center), Roanoke (Virginia Prosthetics & orthotics) and Orlando (Ossur facility, Florida gait lab) . Participants had to visit the study location twice, for approximately 3 hours per visit. First time for the baseline measure and initial fitting and secondly after 3 weeks of accommodation on the Rheo knee XC, performing the same measures as for the baseline. No standard exists for follow up time needed for amputees to adapt to a new prosthesis however, a follow up time of at least 3 weeks is widely used and considered sufficient for functional comparison.

All users used their existing sockets throughout the testing without modifications. One group consisted of 9 previous MPK-magnetorheologic (MPK-MR), Rheo knee II and III, users and the second group of 4 previous MPK-hydraulic knee (MPK-HY), Genium, users. By maintaining alignment and foot choice in the previous Rheo knee group confounding factors could be minimized. The previous MPK-HY was provided with an alignment offset adapter and a consistent foot choice, XC Vari-Flex, at initial fitting. The load line was controlled to be equal prior and post initial fitting. During the initial fitting the MPK-HY users which were new to the XC Vari-Flex had to undergo an evaluation for the foot stiffness as defined by the manufacturer (Ossur ehf). Foot configuration had to be rated acceptable or better with all users that were provided with a XC Vari-Flex.

13 users completed a 3 week evaluation in a multi-center trial with the RHEO KNEE XC at which point they performed Borg Scale CR 10 pre, 6MWT, Borg Scale CR 10 post, L-Test, stair and bicycle evaluation and prosthesis evaluation quesionnaire mobility section) PEQ MS 12/5) on functional ability and prosthesis satisfaction in this order.

The Borg Scale CR 10 is an accepted and reliable psychophysical score which has been used to report on the perceived level of exertion in lower limb amputees. The 6MWT has shown to be a reliable measure in amputees and differentiate among functional levels with a minimum detectable change for unilateral trans-tibial and transfemoral found at 45m. The L-Test is a valid indicator for functional mobility and showed high intraclass correlation, interrater reliability, and minimal bias upon retesting with a moderate correlation to self-reports like the PEQ MS 12/522 which itself is a reliable and valid measure for lower limb amputee assessing psychometric properties.

Ambulating stairs was evaluated as a timed parameter split up in ascending and descending. An observer score/SAI for the gait quality, and a user score/self-report with a 5 point scale (Please rate your ability when using the prosthesis: unable=0, highly difficult=1, moderate difficulty=2, little difficulty=3, no problems=4) similar to the PEQ MS 12/5 scores described by Franchignoni et. al.22 was used. The Rheo Knee XC stair mode can be entered by flexing the hip of the amputated side faster and to a higher degree than in typical walking. The Rheo knee XC will then maintain a flexed position to allow the user to position the foot onto the next stair case. The Genium requires the amputee to stop in front of the stairs and initiate a fast movement into hip-hyperextension to allow the knee to maintain a flexed position. For adapting these two different techniques each user was given 30min training time with instructions to get familiar with the stairs and the operation of the knee in specific location. Equal time was given after initial fitting which was important to the previous MPK-MR knee users who have not used the stair mode before. For the bicycle evaluation the same 5 point scale for the self-report assessment was applied to report on 2 questions: Rate your ability to ride the bicycle and rate your ability to stop the bike with the prosthetic side down.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive ability to understand all instructions and questionnaires in the study;
* Unilateral kneedisartic or transfemoral users fitted to Rheo Knee II,III Genium or X2 or X3
* Willing and able to participate in the study and follow the protocol
* Confident prosthetic users for more than 3 months
* Older than 18 years

Exclusion Criteria:

* 50Kg> body weight > 136Kg
* Users with cognitive impairment
* Users not understanding the function of the knee
* Users not able to charge the battery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2015-08-04 (Actual); Study Completion 2015-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Pratt, M.Sc., Principal Investigator — Ossur Iceland ehf
Locations (4):
- United States (4):
  - Ossur Americas, Florida Gait lab, Orlando, Florida
  - Methodist Rehabilitation Center, Flowood, Mississippi
  - Baker Orthotics & Prosthetics, Fort Worth, Texas
  - Virginia Prosthetics & Orthotics, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hafner BJ, Willingham LL, Buell NC, Allyn KJ, Smith DG. Evaluation of function, performance, and preference as transfemoral amputees transition from mechanical to microprocessor control of the prosthetic knee. Arch Phys Med Rehabil. 2007 Feb;88(2):207-17. doi: 10.1016/j.apmr.2006.10.030. PMID 17270519
- [Background] Starholm IM, Gjovaag T, Mengshoel AM. Energy expenditure of transfemoral amputees walking on a horizontal and tilted treadmill simulating different outdoor walking conditions. Prosthet Orthot Int. 2010 Jun;34(2):184-94. doi: 10.3109/03093640903585016. PMID 20141493
- [Background] Borg G. Psychophysical scaling with applications in physical work and the perception of exertion. Scand J Work Environ Health. 1990;16 Suppl 1:55-8. doi: 10.5271/sjweh.1815. PMID 2345867
- [Background] Gailey RS, Roach KE, Applegate EB, Cho B, Cunniffe B, Licht S, Maguire M, Nash MS. The amputee mobility predictor: an instrument to assess determinants of the lower-limb amputee's ability to ambulate. Arch Phys Med Rehabil. 2002 May;83(5):613-27. doi: 10.1053/apmr.2002.32309. PMID 11994800
- [Background] Deathe AB, Miller WC. The L test of functional mobility: measurement properties of a modified version of the timed "up & go" test designed for people with lower-limb amputations. Phys Ther. 2005 Jul;85(7):626-35. PMID 15982169
- [Background] Franchignoni F, Monticone M, Giordano A, Rocca B. Rasch validation of the Prosthetic Mobility Questionnaire: A new outcome measure for assessing mobility in people with lower limb amputation. J Rehabil Med. 2015 May;47(5):460-5. doi: 10.2340/16501977-1954. PMID 25783231
- [Background] Resnik L, Borgia M. Reliability of outcome measures for people with lower-limb amputations: distinguishing true change from statistical error. Phys Ther. 2011 Apr;91(4):555-65. doi: 10.2522/ptj.20100287. Epub 2011 Feb 10. PMID 21310896
- [Background] Franchignoni F, Giordano A, Ferriero G, Orlandini D, Amoresano A, Perucca L. Measuring mobility in people with lower limb amputation: Rasch analysis of the mobility section of the prosthesis evaluation questionnaire. J Rehabil Med. 2007 Mar;39(2):138-44. doi: 10.2340/16501977-0033. PMID 17351696

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheo Knee XC
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rheo Knee XC
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Weight [Mean (Standard Deviation); unit: Kg] | 82 (17.3)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test (6MWT)
Description: The 6MWT is simply a record of the distance traveled by a given patient at his or her self-selected walking speed over a period of six minutes. All that is required is a stopwatch and a walking corridor or track of known distance. Those administering the test should avoid walking with or in front of test subjects to avoid pacing individuals outside of their self-selected walking speed.
  The outcome of the test is the distance walked in 6 minutes, in meters.
Time Frame: Measured at baseline and after 3 weeks follow up.
Population: The outcome reported was collected at 3 week follow up on the investigational device.
Measure: Mean (Full Range); unit: Meters
Groups:
- Baseline: Measurements on subjects usual prosthesis
Arm/Group | Rheo Knee XC | Baseline
Number analyzed (Participants) | 13 | 13
Meters | 506 [376 to 667] | 428.23 [340 to 590]

ADVERSE EVENTS:
Arm/Group | Rheo Knee XC
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes